CLINICAL TRIAL: NCT00553306
Title: Phase I Study To Evaluate Cellular Adoptive Immunotherapy Using Autologous CD8+ Antigen-Specific T Cell Clones Following Cyclophosphamide Conditioning For Patients With Metastatic Melanoma
Brief Title: Laboratory-Treated T Cells and Aldesleukin After Cyclophosphamide in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2179.00; NCI-2010-01281
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; Interleukins; Cyclophosphamide; Biopsy; Immunohistochemistry; Flow Cytometry; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Beginning 48 hours before T-cell infusion, patients receive cyclophosphamide IV. Patients then receive antigen-specific CD8+ T cells IV alone or with CD4+ T helper clones over 1-2 hours on day 0. Patients also receive aldesleukin subcutaneously twice daily on days 0-13. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: therapeutic autologous lymphocytes; Biological: aldesleukin; Drug: cyclophosphamide; Procedure: biopsy; Other: immunohistochemistry staining method; Other: flow cytometry; Genetic: polymerase chain reaction

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes — Given IV
  Other Names: AL; Autologous Lymphocytes; autologous T cells
Biological: aldesleukin — Given subcutaneously
  Other Names: IL-2; interleukin II; Proleukin; recombinant human interleukin-2; recombinant interleukin-2; TCGF, interleukin
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies
Other: immunohistochemistry staining method — Optional correlative studies
  Other Names: immunohistochemistry
Other: flow cytometry — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR

SUMMARY:
RATIONALE: Laboratory-treated T cells may be able to kill tumor cells when they are put back into the body. Aldesleukin and cyclophosphamide may stimulate the immune system in different ways and stop tumor cells from growing. Giving laboratory-treated T cells together with aldesleukin after cyclophosphamide may be an effective treatment for melanoma.

PURPOSE: This phase I/II trial is studying the side effects of giving laboratory-treated T cells together with aldesleukin after cyclophosphamide and to see how well they work in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and toxicity of cellular adoptive immunotherapy in melanoma patients using autologous CD4+ and CD8+ antigen-specific T cell clones.

II. To evaluate the antitumor effects of CD4+ and CD8+ antigen-specific T cells in patients with metastatic melanoma.

III. To determine the duration of in vivo persistence of adoptively transferred CD8+ antigen-specific T cell clones in the presence or absence of transferred CD4+ T cells.

SECONDARY OBJECTIVES:

I. To assess the in vivo antitumor efficacy of the infused autologous antigen-specific CD4+ T cells.

OUTLINE: This is a phase I study followed by a phase II study.

Beginning 48 hours before T-cell infusion, patients receive cyclophosphamide IV. Patients then receive antigen-specific CD8+ T cells IV alone or with CD4+ T helper clones over 1-2 hours on day 0. Patients also receive aldesleukin subcutaneously twice daily on days 0-13. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up weekly for 8 weeks, and then periodically thereafter.

ELIGIBILITY:
Inclusion

* Histopathologically documented metastatic melanoma
* Karnofsky Performance status of at least 70%
* Expected survival of greater than 16 weeks
* WBC > 2,500/uL (ANC > 1,000 uL)
* Platelet count > 80,000 uL
* HCT > 28%
* Patients whose tumor expresses targeted antigen and restricting allele against which CD4 and CD8 T cell clones can be generated
* No CNS metastasis
* Patient's whose tumor expresses an antigen and HLA type for which both an HLA Class I and HLA Class II epitope are listed, will be eligible for this study
* CD4 and CD8 T cell clones do not necessarily have to target the same antigen to be eligible for the study, it is only necessary that the targeted antigen is expressed by the tumor and its epitope is restricted by an HLA allele expressed by the patient
* Evidence of measurable residual disease by clinical exam or imaging studies

Exclusion

* Current central nervous system metastases; patients with history of CNS metastases that show no current evidence of active disease are eligible
* Patients with active infections or oral temperature > 38.2 C within 72 hours of study entry or systemic infection requiring chronic maintenance or suppressive therapy
* Current treatment with steroids
* Patients who are HIV seropositive (poor CD4 T cell generation due to low CD4 T cell recovery and likely HIV reservoir in stimulator cells used in vitro culture)
* Prognosis less than 6 months
* FOR T CELL INFUSION:
* Pregnant women, nursing mothers of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to entry
* Serum creatinine > 2.0 mg/dL
* Significant hepatic dysfunction (hepatic toxicity >= grade 2 (NCICTC) of whatever origin
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing and those with FEV1 < 60% of normal or DLco (corr for Hgb) < 55% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following: congestive heart failure, clinically significant hypotension, symptoms of coronary artery disease, presence of cardiac arrhythmias on EKG requiring drug therapy
* Ejection fraction < 50% excludes patients
* Current central nervous system metastases; patients with history of CNS metastases that show no current evidence of active disease are eligible
* Serum calcium > 12 mg/dL
* Chemotherapeutic agents (standard or experimental), radiation therapy, or other immunosuppressive therapies less than 4 weeks prior to T cell therapy; patients with bulky disease may undergo 1-2 courses of cytoreductive chemotherapy but treatment will be discontinued at least 4 weeks prior to T cell therapy; patients should have recovered fully from all previous treatment-related toxicities
* History of seizures
* Patients must not be receiving any other experimental drugs within 4 weeks of the initiation of the protocol and must have recovered from all side effects of such therapy
* Patients with >= Grade 2 hepatotoxicity are excluded
* Patients with a history of autoimmune disease requiring active systemic therapy are excluded
* The following agents are not allowed while on study: systemic corticosteroids (except as outlined for management of toxicity of nontransduced CTL), immunotherapy (for example, interleukins, interferons, melanoma vaccines, intravenous immunoglobulin, expanded polyclonal TIL or LAK therapy), pentoxifylline, or other investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity as assessed by NCI CTC version 3.0 | 8 weeks post treatment
Antitumor effects of CD4+ and CD8+ antigen-specific T-cells | 8 weeks post treatment
Duration of in vivo persistence of adoptively transferred CD8+ antigen-specific T cell clones in the presence or absence of transferred CD4+ T cells | 8 weeks post treatment

SECONDARY OUTCOMES:
In vivo antitumor efficacy of the infused autologous antigen-specific CD4+ T cells | 8 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States